CLINICAL TRIAL: NCT01901848
Title: Combined Smoking Cessation and Cognitive Processing Therapy for PTSD
Brief Title: CPT and Smoking Cessation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MHBA-018-12F
Record Dates: First submitted 2013-07-12; First posted 2013-07-17 (Estimated); Results first posted 2018-09-11 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-08

CONDITIONS: Stress Disorders, Post-Traumatic; Smoking
Keywords: Smoking Cessation; Stress Disorders, Post-Traumatic; Psychotherapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Smoking; Smoking Cessation | interventions — Bupropion; Nicotine Replacement Therapy; Nicotine; Nicotine Chewing Gum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- CPT+ICSC (Experimental): This arm includes 12 sessions of combined Cognitive Processing Therapy (CPT) and Integrated Care for Smoking Cessation (ICSC), involvement in smokefreeVET.gov's text messaging program for smoking cessation, Bupropion use, and nicotine replacement therapy.
  Interventions: Behavioral: Cognitive Processing Therapy (CPT); Drug: Bupropion; Drug: nicotine replacement therapy (NRT); Behavioral: Integrated Care for Smoking Cessation (ICSC); Behavioral: smokefreeVET
- ICSC only (Active Comparator): This arm includes 12 sessions of Integrated Care for Smoking Cessation (ICSC), involvement in smokefreeVET.gov's text messaging program for smoking cessation, Bupropion use, and nicotine replacement therapy.
  Interventions: Drug: Bupropion; Drug: nicotine replacement therapy (NRT); Behavioral: Integrated Care for Smoking Cessation (ICSC); Behavioral: smokefreeVET

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy (CPT) — CPT is based on a social cognitive theory of PTSD that includes primary emotional responses to traumatic events such as fear, anger, and sadness, as well as secondary emotions resulting from a patient's faulty interpretations of the traumatic event. CPT addresses PTSD by facilitating affective expression so that affective components of the trauma memory can be altered. In addition, faulty beliefs about the trauma are challenged and modified using Socratic questioning.
  Arms: CPT+ICSC
Drug: Bupropion — Bupropion is an anti-depressant medication that is commonly used in smoking cessation treatment.
  Other Names: Zyban
Drug: nicotine replacement therapy (NRT) — NRT in the form of nicotine patches and an NRT rescue method (e.g., nicotine gum, lozenge, inhaler) will be prescribed for participants for use on/after quit date.
  Other Names: Nicoderm, Nicorette
Behavioral: Integrated Care for Smoking Cessation (ICSC) — ICSC is a manualized treatment for smoking cessation involving six sessions of counseling.
Behavioral: smokefreeVET — SmokefreeVET is a program that was developed by the National Institutes of Health and Department of Veterans Affairs. The program includes a text messaging protocol for reaching out to Veterans who wish to stop smoking.

SUMMARY:
Posttraumatic stress disorder (PTSD) and cigarette smoking are both associated with significant impairment in Veterans and cost to the Veterans' Affairs (VA) system. Though research suggests smoking is linked with PTSD symptoms, existing smoking cessation treatments targeting PTSD smokers do not include PTSD treatment. The purpose of this study is to examine a treatment that combines evidence based treatment for PTSD (cognitive processing therapy, or CPT) with smoking cessation treatment for PTSD and a mobile text messaging program. The study objectives are to evaluate feasibility of the treatment and to examine effectiveness of CPT and smoking cessation treatment combined compared to smoking cessation treatment without CPT. Fifty Veteran smokers with PTSD will participate in fourteen study sessions, ending with the final follow-up session six months after the scheduled quit date.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) and cigarette smoking are both associated with significant impairment in Veterans and cost to the Veterans' Affairs (VA) system. Though naturalistic and laboratory studies suggest smoking is linked with PTSD symptoms, existing smoking cessation treatments targeting PTSD smokers have not utilized standardized, evidence-based PTSD treatment. The most effective smoking cessation approach to date for PTSD smokers, Integrated Care for Smoking Cessation (ICSC), relies on delivery of smoking cessation treatment by the individual's PTSD treatment provider. In a recent trial comparing ICSC to VA specialty Smoking Cessation Clinic care, ICSC produced significantly better prolonged smoking abstinence. However, ICSC was associated with only modest improvements in PTSD symptoms, with no difference between ICSC and smoking cessation treatment alone, suggesting a likely avenue for improving ICSC. The investigators have developed an intervention that combines evidence based treatment for PTSD [cognitive processing therapy (CPT-C)] with evidence based smoking cessation for PTSD [Integrated Care for Smoking Cessation (ICSC)] and a mobile text messaging program. The primary aim of the proposed study is to evaluate the integration of CPT-C and smoking cessation treatment in an individual 12-session PTSD protocol as compared to a protocol including the same smoking cessation treatment for individuals with PTSD, but without CPT-C. This intervention will be evaluated with the following hypotheses:

1. Compared to the smoking cessation alone protocol, the smoking cessation + concurrent CPT-C protocol will result in reduced frequency and intensity of PTSD symptoms.
2. Compared to the smoking cessation alone protocol, the smoking cessation + concurrent CPT-C protocol will result in reduced depressive symptoms.
3. The smoking cessation + concurrent CPT-C protocol will result in decreased smoking rates, relative to published data on VA smoking cessation usual care.
4. Greater PTSD symptom reduction during the smoking cessation + concurrent CPT-C treatment will result in longer duration to smoking lapse and relapse.
5. Exploratory research question: Will candidate genes described earlier predict treatment response in smokers with PTSD?
6. Exploratory research question: Will use of automated text messaging as an adjunct to smoking cessation be feasible, and will it impact quit rates?

The development of a combined CPT-C/ICSC intervention with established empirical support would benefit the many Veterans with PTSD who smoke by providing them with treatment of two pervasive problems with significant associated impairment. In addition, this treatment could substantially reduce the cost of administering two individual treatments separately by administering them in combination.

ELIGIBILITY:
Inclusion Criteria:

* Must be U.S. Veteran
* Smoke at least ten cigarettes a day
* Meet criteria for current PTSD
* Speak and write fluent conversational English
* Be between 18 and 65 years of age
* Be willing to attempt smoking cessation
* Must have access to a phone capable of receiving text messages

Exclusion Criteria:

* Not stable on medications for the study period
* History of myocardial infarction in the past 6 months
* Contraindication to NRT and inability to get medical clearance from primary care provider
* Use of other forms of nicotine such as cigars, pipes, or chewing tobacco.
* Pregnancy
* Inability to complete study measures and tasks independently
* Dementia or other brain disorder, schizophrenia, current manic syndrome, or substance abuse/dependence in the preceding 3 months.
* Currently receiving trauma-focused psychotherapy.
* Currently living in court-ordered residential substance abuse treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2013-12-11 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric A Dedert, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dedert EA, Resick PA, Dennis PA, Wilson SM, Moore SD, Beckham JC. Pilot Trial of a Combined Cognitive Processing Therapy and Smoking Cessation Treatment. J Addict Med. 2019 Jul/Aug;13(4):322-330. doi: 10.1097/ADM.0000000000000502. PMID 30664539

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 69 participants consented before the screening session. Nineteen were excluded, and 50 were randomized. As a result, there were 69 who consented, but only 50 are included in the flow diagram for the trial.
Groups:
- CPT+ICSC: This arm includes 12 sessions of combined Cognitive Processing Therapy (CPT) and Integrated Care for Smoking Cessation (ICSC), involvement in smokefreeVET.gov's text messaging program for smoking cessation, Bupropion use, and nicotine replacement therapy.
  Cognitive Processing Therapy (CPT): CPT is based on a social cognitive theory of PTSD that includes primary emotional responses to traumatic events such as fear, anger, and sadness, as well as secondary emotions resulting from a patient's faulty interpretations of the traumatic event. CPT addresses PTSD by facilitating affective expression so that affective components of the trauma memory can be altered. In addition, faulty beliefs about the trauma are challenged and modified using Socratic questioning.
  Bupropion: Bupropion is an anti-depressant medication that is commonly used in smoking cessation treatment.
  nicotine replacement therapy (NRT): NRT in the form of nicotine patches and an NRT rescue method (e.g., nicotine gum,
- Present-focused ICSC: This arm includes 12 sessions of Integrated Care for Smoking Cessation (ICSC), involvement in smokefreeVET.gov's text messaging program for smoking cessation, Bupropion use, and nicotine replacement therapy.
  Bupropion: Bupropion is an anti-depressant medication that is commonly used in smoking cessation treatment.
  nicotine replacement therapy (NRT): NRT in the form of nicotine patches and an NRT rescue method (e.g., nicotine gum, lozenge, inhaler) will be prescribed for participants for use on/after quit date.
  Integrated Care for Smoking Cessation (ICSC): ICSC is a manualized treatment for smoking cessation involving six sessions of counseling.
  smokefreeVET: SmokefreeVET is a program that was developed by the National Institutes of Health and Department of Veterans Affairs. The program includes a text messaging protocol for reaching out to Veterans who wish to stop smoking.
Period: Randomized and Treated
Arm/Group | CPT+ICSC | Present-focused ICSC
Started | 25 | 25
Completed | 22 (Ten cases were practice cases used to establish fidelity to CPT, and were removed from analyses.) | 19
Not Completed | 3 | 6
Not completed — Lost to Follow-up | 3 | 6
Period: Removed From Analyses
Arm/Group | CPT+ICSC | Present-focused ICSC
Started | 22 | 19
Completed | 12 | 19
Not Completed | 10 | 0
Not completed — CPT practice cases to establish fidelity | 10 | 0

BASELINE CHARACTERISTICS:
Population: Because primary analyses used maximum likelihood to address missing data, participants who were lost to follow-up (n = 3 in CPT+ICSC group, n = 6 in ICSC group) were included in primary analyses.
Groups:
- CPT+ICSC: This arm includes 12 sessions of combined Cognitive Processing Therapy (CPT) and Integrated Care for Smoking Cessation (ICSC), involvement in smokefreeVET.gov's text messaging program for smoking cessation, Bupropion use, and nicotine replacement therapy.
  Cognitive Processing Therapy (CPT): In CPT, faulty beliefs about the trauma are challenged and modified using Socratic questioning.
  Bupropion: Bupropion is an anti-depressant medication that is commonly used in smoking cessation treatment.
  nicotine replacement therapy (NRT): NRT in the form of nicotine patches and an NRT rescue method (e.g., nicotine gum,
- Total: Total of all reporting groups
Arm/Group | CPT+ICSC | Present-focused ICSC | Total
Number analyzed (Participants) | 15 | 25 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.1 (10.8) | 53.3 (10.8) | 49.5 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 6 | 7
  Male | 14 | 19 | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 9 | 14 | 23
  Caucasian, not Hispanic | 3 | 7 | 10
  Hispanic | 2 | 0 | 2
  Multiple Races | 1 | 4 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 25 | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Self-report 7-day Point Prevalence Smoking Abstinence at 6-month Follow-up.
Description: 7-day point prevalence abstinence is defined as participant reporting no smoking occasions in the 7 days preceding the 6-month follow-up appointment. The 6-month follow-up occurs 6 months after the initial scheduled quit date.
Time Frame: 6-month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | CPT+ICSC | Present-focused ICSC
Number analyzed (Participants) | 15 | 25
Participants | 2 | 8

2. Primary Outcome: Number of Participants Who Self-reported 7-day Point Prevalence Smoking Abstinence as Bioverified by Breath Carbon Monoxide < 4 Parts Per Million.
Description: Self-reported 7-day point prevalence smoking abstinence was bioverified by breath carbon monoxide level of < 4 parts per million at the 6-month follow-up.
Time Frame: 6-month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | CPT+ICSC | Present-focused ICSC
Number analyzed (Participants) | 15 | 25
Participants | 2 | 4

ADVERSE EVENTS:
Time Frame: For participants in the CPT+ICSC condition, adverse event data were collected for approximately 8 months. For participants in the ICSC condition, adverse event data were collected for up to 12 months.
Description: n/a; clinicaltrials.gov definition used.
Arm/Group | CPT+ICSC | Present-focused ICSC
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/15 | 2/25
Other Adverse Events (participants affected / at risk) | 5/15 | 4/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CPT+ICSC (N=15) | Present-focused ICSC (N=25)
Hospitalization due to alcohol intoxication/withdrawal (Psychiatric disorders) | 0 (0) | 1 (1) — Due to pre-existing substance use disorder; not study-related
Hospitalization due to antibiotic reaction (General disorders) | 0 (0) | 1 (1) — Pt. was given antibiotics for bee sting, had negative reaction to prescribed meds. Not study related.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CPT+ICSC (N=15) | Present-focused ICSC (N=25)
Increased anxiety (Psychiatric disorders) | 0 (0) | 2 (2) — Reported increased anxiety and irritability. Potentially study-related, as anxiety is known feature of PTSD.
Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) — Reported increased congestion. Possible study related, because is side effect of quitting smoking.
Cervicalgia (Reproductive system and breast disorders) | 1 (1) | 0 (0) — Pre-existing condition, not study related
Stomach pain/flank pain (Gastrointestinal disorders) | 0 (0) | 2 (2) — Not study related
Flu-like symptoms (General disorders) | 1 (1) | 0 (0) — Not study related
Increased arthritis symptoms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Due to pre-existing condition, not study-related
Itchiness/skin irritation at site of nicotine patch (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Itchiness/skin irritation is a known side effect of nicotine patch use.
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) — Nausea is known potential side effect of nicotine replacement therapies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-01-09): https://cdn.clinicaltrials.gov/large-docs/48/NCT01901848/Prot_SAP_ICF_000.pdf